CLINICAL TRIAL: NCT04955041
Title: Effectiveness of T2* MRI in Predicting Prognosis in Patients With Cervical Spondylotic Myelopathy (CSM)
Brief Title: Effectiveness of T2* MRI in Cervical Spondylotic Myelopathy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020317
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2020-07

CONDITIONS: Cervical Spondylotic Myelopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mild CSM: preoperative modified Japanese Orthopedic Association (mJOA) score ≥15
  Interventions: Other: MRI
- moderate CSM: preoperative mJOA score 13~14
  Interventions: Other: MRI
- severe CSM: preoperative mJOA score ≤12
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — T2* MRI

SUMMARY:
Utilization of T2* MRI in predicting prognosis in patients with cervical spondylotic myelopathy (CSM)

DETAILED DESCRIPTION:
Cervical spondylotic myelopathy (CSM), an age-related degenerative disease that is common worldwide, is mainly caused by compression of the spinal cord and may possibly lead to disability. Surgery to reduce direct compression of the spinal cord might alleviate disease progression; due to individual differences, some patients do not benefit from surgery. Prognostic prediction is important because it affects subsequent treatment decision making. Currently, prognosis is generally based on magnetic resonance imaging (MRI) with a detailed macrostructural evaluation of the spinal cord. Unfortunately, the use of conventional MRI indicators (e.g., increased intensity signal [ISI]) to predict CSM outcomes has been controversial because of their subjectivity or the insufficient information contained therein.

A new biomarker, T2* MRI gray matter to white matter signal intensity ratio (GM/WM), is associated with demyelination and gliosis. Previous studies have shown that patients with CSM can have T2* MRI WM / GM changes at the early stage of disease, and the WM / GM value is increased, which is significantly higher than that of normal people, and is related to the spinal cord function score. However, the correlation between this index and long-term prognosis remains to be studied.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with CSM and operated on by one senior orthopedist
* available preoperative MRI results
* high-quality image data with no motion artifacts
* available preoperative and long-term follow-up (≥1 years) mJOA score

Exclusion Criteria:

* prior head or neck surgery
* a history of notable additional diseases (spinal cord tumor, multiple sclerosis, syringomyelia, spinal cord injury, or motor neuron disease).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients came from Peking University Third Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-01 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Improvement of neurologic function | at follow-up time (≥1 years)
  Postoperative modified Japanese Orthopaedic Association (mJOA) at follow-up time

CONTACTS AND LOCATIONS:
Overall Officials: Huishu Yuan, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No
No.